CLINICAL TRIAL: NCT07324226
Title: Effects of Combined Heat Application and Acupressure to the Carotid Artery Region on Cerebral Blood Flow in Healthy Adults: An Investigator-Initiated, Single-Group, Single-Center, Prospective Case Study
Brief Title: Effects of Combined Heat Application and Acupressure to the Carotid Artery Region on Cerebral Blood Flow in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-2025-010
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects/Volunteers
Keywords: Carotid artery; Heat application; SPECT imaging; Acupressure Combined heat and acupressure; Cerebral blood flow; Single-group prospective study; Single-center study
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined heat and acupressure (Experimental): Combined heat and acupressure
  Interventions: Device: Combined heat and acupressure

INTERVENTIONS:
Device: Combined heat and acupressure — Press the start button to activate the automatic mode. When the start button is pressed, the device operates for approximately 40 minutes.
  When the start button is pressed, acupressure massage is performed with a single back-and-forth cycle from acupressure bar No. 1 to No. 18.
  The device then performs back-and-forth acupressure massage between acupressure bars No. 18 and No. 13 for the remaining time.
  After operating for 40 minutes in automatic mode, the mattress heating unit, the acupressure bar heating unit, and the acupressure bar movement are all turned off.
  1. Press the shoulder button. The acupressure bar operates in the neck-to-shoulder section (acupressure bars No. 1 to 6), and both the mattress heating unit and the acupressure bar heating unit are activated.
  2. After operating for 20 minutes in manual mode, the mattress heating unit, the acupressure bar heating unit, and the acupressure bar movement are turned off.

SUMMARY:
The aim of this study is to investigate the effects of combined heat application and acupressure to the carotid artery region on cerebral blood flow in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 65 years.
* Individuals with no history of cerebrovascular, cardiovascular, or neurological diseases.
* Individuals who have signed the informed consent form and voluntarily agreed to participate in the study

Exclusion Criteria:

* Individuals with a history of cerebrovascular, cardiovascular, or neurological diseases (e.g., stroke, angina, epilepsy).

Individuals currently taking medications that may affect cerebral blood flow (such as antihypertensive agents or antidepressants).

Individuals with skin diseases or lesions that make it difficult to apply heat or acupressure devices to the carotid artery region, and individuals who are pregnant or breastfeeding.

Individuals with a history of seizures.

Individuals who have participated in clinical studies two or more times in the same year, or who have participated in another clinical study within the past 6 months.

Individuals who, in the judgment of the principal investigator or sub-investigator, have clinically significant findings that make them unsuitable for participation in this study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A SPECT CT brain scan | In the post-SPECT protocol, the radiopharmaceutical will be administered at 5 minutes (n=3), 10 minutes (n=3), and 20 minutes (n=3) after the start of image acquisition.
  Cerebral blood flow change rate analysis: For each participant, the percentage change in cerebral blood flow (CBF) observed on SPECT imaging compared with the baseline time point will be quantitatively analyzed at the following three time points.
  Radiopharmaceutical injection reference times: 5 minutes, 10 minutes, and 20 minutes after injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab lab, Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared due to protection of participants' personal infand regulatory restrictions of our hospital.